CLINICAL TRIAL: NCT01622725
Title: Recurrence Rate After Primary and Secondary Ventral Hernia Repair Using Long-term Resorbable Versus Non-resorbable Large Pore Synthetic Mesh.
Brief Title: Primary and Secondary Ventral Hernia Repair Using Long-term Resorbable Versus Non-resorbable Large Pore Synthetic Mesh.
Acronym: TIGR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Ghent (Other)
Collaborators: Novus Scientific (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2012/223
Record Dates: First submitted 2012-06-15; First posted 2012-06-19 (Estimated); Last update posted 2024-06-03 (Actual); Status verified 2024-05

CONDITIONS: Primary and Secondary Ventral Hernia
Keywords: ventral hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Resorbable mesh (Experimental): Long-term resorbable mesh implanted to treat primary and secondary ventral hernia.
  Interventions: Procedure: Placing the resorbable mesh
- Non-resorbable mesh (Active Comparator): Non-resorbable synthetic mesh implanted to treat primary and secondary ventral hernia.
  Interventions: Procedure: Non-resorbable synthetic mesh.

INTERVENTIONS:
Procedure: Placing the resorbable mesh — Surgery for primary and secondary ventral hernia repair with placing of resorbable mesh.
  Arms: Resorbable mesh
Procedure: Non-resorbable synthetic mesh. — Surgery for primary and secondary ventral hernia repair with placing of non-resorbable synthetic mesh.
  Arms: Non-resorbable mesh

SUMMARY:
Since abdominal wall hernia repair is currently performed with the use of a mesh, side effects associated with the mesh are frequently reported during long term follow-up. These side effects are related to shrinkage of the mesh, adhesions to the bowl, pain, and inflammation of the skin and bowl. To reduce or prevent these effects, a fully resorbing mesh has been developed, which provides sufficient support and strength to allow efficient recovery of the abdominal wall, but also disappear from your body in three years time, so that you no longer have any synthetic material in your body. Previous resorbing meshes also disappeared but over a much shorter period of time, so that the hernia was insufficiently healed, with recurrence as a result.

The TIGR™ mesh (the resorbable mesh used in the study) is in principle a synthetic mesh, made of two commonly used polymers, however it will retain 50% of its initial strength after six months. This in theory is enough to provide support of the collagen healing process during the initial wound-healing phase, but also to support the transition of initial collagen to functional collagen.

The aim of this study is to compare TIGR™ with large pore mesh used in the repair of the anterior abdominal wall repair (incisional hernia, umbilical hernia, etc..Inguinal hernias are not part of the study).

Therefore the patients will be divided into two groups, one group will be treated with a resorbing mesh, the other group will be treated with a permanent mesh. Otherwise there will be no difference in the medication or the surgical techniques used.

ELIGIBILITY:
Inclusion Criteria:

* Primary and secondary ventral hernia

  * less than 20 cm in length
  * less than 6 cm in width

Exclusion Criteria:

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2013-02 (Actual); Primary Completion 2021-08-01 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Recurrence rate at 3 years post-surgery. | 3 years post-surgery
  Clinical evaluation and ultrasound evaluation after 3 years post-surgery.

SECONDARY OUTCOMES:
Wound Morbidity 4 weeks post-surgery. | 4 weeks post-surgery
Pain and discomfort after 1 year post-surgery. | After 1 year post-surgery
Pain and discomfort after 3 years post-surgery. | After 3 years post-surgery
Recurrence rate by clinical examination 1 year post-surgery. | After 1 year post-surgery.
  Clinical Examination to determine the recurrence rate.

CONTACTS AND LOCATIONS:
Overall Officials: Frederik Berrevoet, MD, PhD, Principal Investigator — University Hospital, Ghent
Locations (6):
- Belgium (2):
  - Ghent University Hospital, Ghent
  - University Hospital Leuven, Leuven
- University of Copenhagen, Copenhagen, Denmark
- ul Jagalskiego, Wejherowo, Poland
- Hospital de 12 Octobre, Madrid, Spain
- Royal Infirmary of Edinburgh, Edinburgh, United Kingdom

REFERENCES:
- See also: Related Info — http://www.uzgent.be